CLINICAL TRIAL: NCT05782413
Title: Effect of Mechanical Vestibular Stimulation On Hand Function In Children With Hemiparetic Cerebral Palsy
Brief Title: Effect of Mechanical Vestibular Stimulation On Hand Function In Hemiparetic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Mohamed Abd El Haleem Ghoniem (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed Abd El Haleem Ghoniem, Principal Investigator, faculty of physical therapy, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EG, KFS lab 2 Research
Record Dates: First submitted 2023-02-24; First posted 2023-03-23 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The child will receive a design exercise program. The therapy was based on the principles of NDTBobath neurodevelopmental therapy.
  Interventions: Other: The design exercise program
- Group B (Experimental): The child will receive a design exercise program for 45 min then mechanical vestibular exercise for 15 mins.
  Interventions: Other: mechanical vestibular stimulation; Other: The design exercise program

INTERVENTIONS:
Other: mechanical vestibular stimulation — Device produces mechanical vestibular stimulation. The child was placed in a sitting position on the swing and his hands grasping the ropes at the sides then the therapist stood behind him and begin pushing the platform in fast and jerky movements in back and front, side to side, and in spinning directions with the child trying to maintain his balance in all different directions.
  Arms: Group B
Other: The design exercise program — A selected therapeutic exercises program was based on the principles of NDTBobath neurodevelopmental therapy, which is effective in controlling spasticity in children with cerebral palsy and improving motor function.
  i. Preparation of structures and mobilizations of the scapula, shoulder joint, and chest according to the NDT-Bobath concept ii. Exercises to increase shoulder mobility and elbow joint extension. iii. Fine motor skill exercises, wrist, and hand

SUMMARY:
The current study will be directed to determine the effect of mechanical vestibular stimulation on fine motor skills and pinch strength in children with hemiparesis. Hemiplegic cerebral palsy causes problems with contraction, sensation, and muscular strength in the upper limbs, and its effective use of muscles for reaching, grasping, releasing, and manipulating objects is often compromised

ELIGIBILITY:
Inclusion Criteria:

* Children will be included in the study if they fulfil the following criteria:

  1. Diagnosed with hemiparetic cerebral palsy.
  2. Age ranged from 4 to 6 years.
  3. Children with spasticity grades ranged from 1 to 1+ according to Modified Ashworth Scale
  4. Both genders will be included.
  5. The child will be able to follow verbal commands and instructions.

Exclusion Criteria:

* Children will be excluded from the study if:

  1. Any congenital or developmental disorders in addition to hemiplegia cerebral palsy.
  2. Current hospitalization for urgent medical reasons.
  3. Severe mental retardation.
  4. Children having visual or auditory defects.
  5. Children who had Botox application to the upper extremity in the past 6 months or had undergone a previous surgical intervention to the wrist and hand.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
fine motor skills | 3 month
  We will use Peabody Developmental Motor Scale (PDMS-2) to measure visual motor integration, grasp and fine motor.
pinch strength | 3 month
  We will use Hand Dynamometer to measure pinch strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided